CLINICAL TRIAL: NCT03342222
Title: Multi-center, Randomized, Open, Parallel, Noninferiority Clinical Trial to Evaluate the Safety and Effectiveness of PEEK Interference Screws in Anterior Cruciate Ligament Reconstruction
Brief Title: The Safety and Effectiveness of PEEK Interference Screws in Anterior Cruciate Ligament Reconstruction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Collaborators: Rejoin Hangzhou Martins Medical Equipment Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Hongbin Lu, Porfessor, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMST-01
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: PEEK Interference Screw; Fixation; Anterior Cruciate Ligament Reconstruction
Keywords: PEEK Interference Screw; Fixation; Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK Interference Screws (Experimental): PEEK Interference Screws provided by Ruijin Hangzhou Martins Medical Equipment Co., Ltd.
  Interventions: Device: Interference Screws
- Biosure PK interference screw (Active Comparator): Biosure PK interference screw from Smith & Nephew plc.
  Interventions: Device: Interference Screws

INTERVENTIONS:
Device: Interference Screws — tibial fixation for ACL reconstruction

SUMMARY:
Anterior cruciate ligament (ACL) rupture is one of the most common injuries in sports medicine. ACL reconstructions are usually performed to restore the stability of knee joint and prevent the secondary meniscal and chondral lesions.

120 Subjects with ACL injury were randomly assigned to two groups for ACL reconstruction.Group one: tibial fixation with PEEK Interference Screws (Rejoin Hangzhou Martins Medical Equipment Co., Ltd.);Group two: tibial fixation with Biosure PK interference screw (Smith & Nephew plc). The subjects will be followed by 12 months after surgery for evaluations.Outcome measures included Lysholm score,IKDC, ADT,Lachman.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily sign the informed consent form; Between the ages of 18 and 75; Positive ADT and positive Lachman test. Unilateral anterior cruciate ligament is confirmed by MRI (without posterior cruciate ligament injury or reconstruction); Tolerated for anterior cruciate ligament reconstruction surgery; Normal contralateral knee

Exclusion Criteria:

1. Do not meet the diagnostic criteria of anterior cruciate ligament injury;
2. With posterior cruciate ligament fracture at the same time;
3. X-ray showed a significant degeneration of the knee (more than four degrees of cartilage injury);
4. Knee flexion less than 90 degree;
5. Abnormal body anatomy;
6. Pregnant, breast-feeding or subjects who plan to become pregnant;
7. Serious osteoporosis, malignant tumors;
8. Allergic to implant materials;
9. Patients with severe malnutrition who can not tolerate surgery;
10. Severe coagulopathy, such as hemophilia;
11. Immunodeficiency diseases, including those requiring long-term use of immunosuppressive agents;
12. The injured knee has a wide range of skin diseases;
13. Serious obese patients (BMI> 35);
14. Patients with severe mental illness can not cooperate with postoperative rehabilitation and patients with severe cardiopulmonary disease can not tolerate surgery;
15. Ipsilateral lower extremity received surgery within the past year;
16. Has participated in any other clinical trial in the past three months;
17. Can not comply with the requirements of the study;
18. Those who the investigator thinks they are inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-11-20 (Estimated); Study Completion 2019-11-20 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with Lysholm score more than 70 score | 12 month

SECONDARY OUTCOMES:
Lysholm score | 1month; 3month; 6 month; 12 month
IKDC | 1month; 3month; 6 month; 12 month
Anterior drawer test | 1month; 3month; 6 month; 12 month
Lachman test | 1month; 3month; 6 month; 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No